CLINICAL TRIAL: NCT00822458
Title: A Phase I Pharmacokinetic and Safety Study in Children With Recurrent or Refractory Medulloblastoma to Identify a Pharmacokinetic Based Dose for GDC-0449
Brief Title: GDC-0449 in Treating Young Patients With Medulloblastoma That is Recurrent or Did Not Respond to Previous Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01180; NCI-2009-01180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000631677; PBTC-025 (Other: Pediatric Brain Tumor Consortium); PBTC-025 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Childhood Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — HhAntag691

ARMS (1):
- Arm I (Experimental): Patients receive oral hedgehog antagonist GDC-0449 once daily on days 1 and 4-28 in course 1 and on days 1-28 in all subsequent courses. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Blood samples are collected periodically for pharmacokinetic studies. Archival tumor tissue samples are collected and analyzed for the expression of genes that activate the SHH (e.g., Gli1, Gli2, SFRP1, ATOH1, and PTCH2) or WNT (e.g., DKK2 and DKK4) cell signal pathways by in situ hybridization and reverse transcriptase real time-PCR.
  Interventions: Drug: vismodegib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: vismodegib — Given orally
  Other Names: Erivedge; GDC-0449; Hedgehog antagonist GDC-0449
Other: laboratory biomarker analysis
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of GDC-0449 in treating young patients with medulloblastoma that is recurrent or did not respond to previous treatment. GDC-0449 may be effective in treating young patients with medulloblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the safety and pharmacokinetics of a daily dose of hedgehog antagonist GDC-0449 using the available formulation in pediatric patients with recurrent or refractory medulloblastoma.

SECONDARY OBJECTIVES:

I. To document and describe toxicities associated with this drug in these patients.

II. To characterize the pharmacokinetics of this drug in these patients. III. To document preliminary antitumor activity of this drug in these patients. IV. To document pathologic and genomic methods to identify CNS tumors with activation of the PTCH/SHH pathway.

OUTLINE: This is a multicenter study.

Patients receive oral hedgehog antagonist GDC-0449 once daily on days 1 and 4-28 in course 1 and on days 1-28 in all subsequent courses. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic studies. Archival tumor tissue samples are collected and analyzed for the expression of genes that activate the SHH (e.g., Gli1, Gli2, SFRP1, ATOH1, and PTCH2) or WNT (e.g., DKK2 and DKK4) cell signal pathways by in situ hybridization and reverse transcriptase real time-PCR.

After completion of study therapy, patients are followed for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed medulloblastoma, including posterior fossa primitive neuroectodermal tumor (PNET)
* Recurrent, progressive, or refractory to standard therapy
* No known curative therapy exists
* Neurological deficits allowed provided they are stable for ≥ 1 week prior to study entry
* No atypical teratoid/rhabdoid tumor or supratentorial PNET
* Karnofsky performance status (PS) 60-100% (for patients > 16 years of age) OR Lansky PS 60-100% (for patients ≤ 16 years of age)
* ANC ≥ 1,000/μL*
* Platelet count ≥ 100,000/μL (transfusion independent)*
* Hemoglobin ≥ 8.0 g/dL (RBC transfusion allowed)*
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age as follows:

  * ≤ 0.8 mg/dL (for patients ≤ 5 years of age)
  * ≤ 1.0 mg/dL (for patients 6 to 10 years of age)
  * ≤ 1.2 mg/dL (for patients 11 to 15 years of age)
  * ≤ 1.5 mg/dL (for patients > 15 years of age)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* ALT/AST ≤ 2.5 times ULN for age
* Serum albumin ≥ 2.5 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use 2 effective methods of contraception during and for 12 months following study treatment
* Fertile male patients must use effective barrier contraception during and for 12 months following study treatment
* Body surface area > 0.67 m^2 and ≤ 2.5 m^2
* Able to swallow capsules
* No malabsorption syndrome or other condition that would interfere with enteral absorption
* No history of congestive heart failure
* No history of ventricular arrhythmia requiring medication
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia, defined as less than the lower limit of normal despite adequate electrolyte supplementation
* No clinically important history of liver disease, including viral hepatitis or cirrhosis
* No concurrent clinically significant unrelated systemic illness (e.g., serious infection) or significant cardiac, pulmonary, hepatic, or other organ dysfunction that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results

  * NOTE: * In the absence of bone marrow involvement
* Recovered from prior treatment-related toxicity
* At least 3 months since prior craniospinal radiotherapy (at doses ≥ 23 Gy)
* At least 8 weeks since prior local radiotherapy to primary tumor
* At least 2 weeks since prior focal radiotherapy to symptomatic metastatic sites
* More than 4 weeks since prior myelosuppressive chemotherapy or immunotherapy (6 weeks for nitrosoureas)
* More than 1 week since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or erythropoietin)
* No other concurrent anticancer or investigational drug therapy
* Concurrent dexamethasone allowed provided dosage is stable or decreasing for ≥ 1 week prior to study entry

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean steady-state total (protein bound and non-protein bound) GDC-0449 plasma concentrations (Css) | 21 days
  95% confidence interval estimates for 2 doses compared.
Pharmacokinetics of GDC-0449, including the elimination rate constant and terminal half life | Up to 3 months after completion of study treatment
  We will study two BSA defined strata.

SECONDARY OUTCOMES:
Tumor responses | Up to 30 days after completion of study treatment
  Descriptive statistics will be provided describing tumor responses.
Progression-free survival | Up to 30 days after completion of study treatment
  Kaplan-Meier estimates of the distribution of progression-free survival (PFS) will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (9):
- United States (9):
  - UCSF-Mount Zion, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas